#### **Cover Page**

## **Participation Consent Form**

Study Title: Unilateral Strength Training and Mirror Therapy for Patients with Chronic

#### Stroke. A Pilot Randomised Controlled

**Trial** Document creation date: July 12th 2015

NCT number [not yet assigned].

Identifiers: [NCT ID not yet assigned]

### **Participation Consent Form**

# Unilateral Strength Training and Mirror Therapy for Patients with Chronic Stroke. A Pilot Randomised Controlled Trial

| 1. | I confirm that I have received a copy of the Information Sheet for the above study. I have read it and I understand it. I have received an explanation of the nature and purpose of the study and what my involvement will be. |
|---|---|
| 2. | I have had time to consider whether to take part in this study and I have had the opportunity to ask questions. |
| 3. | I understand that my participation is voluntary and that I can decide to opt out of the research at any time. |
| 4. | I understand that all information gathered about me during this study will be treated with full confidentiality. |
| 5. | I agree to the video recording of training sessions and understand that all recordings will be kept confidential. |
| 6. | I agree to take part in the above study. |

Date

Signature

Name of patient